CLINICAL TRIAL: NCT04043078
Title: Exercise In Critical Limb Ischaemia Patients Having Surgery
Brief Title: Exercise In Critical Limb Ischaemia Patients Having Surgery Proof of Concept
Acronym: EXERCISE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hull University Teaching Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: R2372
Record Dates: First submitted 2019-07-31; First posted 2019-08-02 (Actual); Last update posted 2020-08-31 (Actual); Status verified 2020-08

CONDITIONS: Critical Limb Ischemia
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise (Other): Exercise and respiratory muscle training before surgery
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — The exercise regime will include daily upper limb aerobic (hand bike) and inspiratory muscle training (POWERbreathe) and upper body strength training every second day until discharge.

SUMMARY:
Patients with critical limb ischaemia (CLI) are at risk of losing their limb and/or life and therefore have no option but to undergo bypass or amputation surgery. This presents a major physical challenge to the body and patients with low fitness will struggle to overcome the effects of the surgical trauma. Currently there is a high risk of a poorer outcome for CLI patients than with most other surgical procedures, as demonstrated by high rates of complications (20-46%) and 30 day mortality (7.5-13.5%). Up to 30% of people will die within the first year. Exercise and respiratory muscle training, before surgery, has shown a reduction in complications in other surgical specialties.

Around 50% of CLI patients present as an emergency, meaning training before admission is not feasible, so the Investigator proposes to see if training during the hospital stay will aid a better recovery. However, as this has not been done in vascular surgical patients the investigator needs to initially test if this intervention is possible in this patient group in an acute hospital setting.The aim of this proof of concept single cohort study is to assess whether an exercise intervention, started on hospital admission and continued post-surgery, for the duration of the hospital admission, is safe, acceptable, well tolerated and feasible to run in an acute ward setting.

The exercise regime will include daily upper limb aerobic (hand bike) and inspiratory muscle training (POWERbreathe) and upper body strength training every second day until discharge. The Investigator will assess safety by recording adverse events and acceptability by adherence to exercise programme and qualitative interviews. The Investigator will evaluate processes and completeness of data collection and describe before and after measures of physical fitness.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old or over
2. Willing to participate and able to give written informed consent
3. Clinical diagnosis of critical limb ischaemia or Fontaine Class III-IV or Rutherford Class 4-6
4. Admitted to the vascular surgical ward for lower limb surgery

Exclusion Criteria:

1. Patients presenting who have diabetes are presenting with acute limb ischaemia with no history of PAD
2. Cognitive Impairment as demonstrated by not being able to safely follow instructions.
3. Unable to understand or read English
4. Absolute contraindications to exercise including:-

   * Acute MI
   * Ongoing unstable angina
   * Uncontrolled cardiac arrhythmia with hemodynamic compromise
   * Active endocarditis
   * Symptomatic severe aortic stenosis
   * Decompensated heart failure
   * Acute pulmonary embolism, pulmonary infarction, or deep vein thrombosis
   * Acute myocarditis or pericarditis
   * Acute aortic dissection
5. Physical disability that precludes safe and adequate exercise as determined by the clinical team
6. Contraindications to IMT including:-

   * A history of spontaneous pneumothrorax (ie not due to traumatic injury)
   * A pneumothorax due to traumatic injury that has not fully healed
   * A burst eardrum that has not fully healed or any other condition of the eardrum
   * Unstable asthma and abnormally low perception of dyspnoea

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-08-03 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Primary (Mortality) | 30 days
  Mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Hull University Teaching Hospitals NHS Trust, Hull, United Kingdom

IPD SHARING:
Plan to Share IPD: No